CLINICAL TRIAL: NCT00053547
Title: Safety and Effectiveness of Zemplar Injection in Decreasing iPTH Levels in Pediatric ESRD Subjects on Hemodialysis
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Abbott (Industry)
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: 2001-022
Record Dates: First submitted 2003-01-30; First posted 2003-02-03 (Estimated); Last update posted 2006-08-02 (Estimated); Status verified 2006-07

CONDITIONS: Secondary Hyperparathyroidism; End Stage Renal Disease
MeSH Terms: conditions — Hyperparathyroidism, Secondary; Kidney Failure, Chronic | interventions — paricalcitol

INTERVENTIONS:
Drug: paricalcitol injection

SUMMARY:
The purpose of this study is to see if Zemplar, a vitamin D medication, safely and effectively decreases parathyroid hormone in children ages 2-20 with End Stage Renal Disease.

ELIGIBILITY:
Subjects ages 2-20 with ESRD on hemodialysis with Secondary hyperparathyroidism

Ages: 2 Years to 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 28
Dates: Start 2002-01

PRIMARY OUTCOMES:
Proportion of subjects achieving at least a 30% decrease from baseline iPTH sustained for at least two consecutive iPTH measurements.

SECONDARY OUTCOMES:
Proportion of subjects in each group who achieve two consecutive iPTH values below 300 pg/mL.

CONTACTS AND LOCATIONS:
Overall Officials: Laura Williams, M.D., Study Director — Abbott
Locations (6):
- United States (6):
  - Stanford University Medical Center, Stanford, California
  - Miami Children's Hospital, Miami, Florida
  - The Children's Hospital of Buffalo, Buffalo, New York
  - Texas Children's Hospital, Houston, Texas
  - University of Texas at Houston, Houston, Texas
  - Medical College of Wisconsin, Milwaukee, Wisconsin